CLINICAL TRIAL: NCT00957398
Title: Comparing of the Gastrointestinal Motility in Irritable Bowel Syndrome (IBS) Patients With Healthy Volunteers Using Magnetic Tracking System (MTS)
Brief Title: Comparing of the Gastrointestinal Motility in Irritable Bowel Syndrome (IBS) Patients With Healthy Volunteers
Status: Terminated | Type: Observational
Why Stopped: Not possible to include patients.
Sponsor: University of Aarhus (Other)
Responsible Party: Principal Investigator, Janne Ladefoged Fassov, PhD student, University of Aarhus
Other Study IDs: 20090009,JLF
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2012-05-10 (Estimated); Status verified 2012-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable Bowel Syndrome; Irritable Bowel Syndrome subgroups; Motility
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- IBS-D: 12 IBS-D patients who will all undergo MTS.
- IBS-C: 12 IBS-C patients who will all undergo MTS.

SUMMARY:
The hypothesis of the study is that the motility of the small intestine and the colon will alter according to the subtype of the irritable bowel syndrome (IBS) patient.

IBS is currently classified into following subtypes:

* Diarrhoea-IBS (IBS-D)
* Constipation-IBS (IBS-C)
* Mixed-IBS (IBS-M)
* Unsubtyped-IBS (IBS-U)

according to the Bristol scale.

Magnetic Tracking System (MTS) is a new minimal invasive technic that allows motility studies of the whole human gastrointestinal tract.

The magnetic cylindrical pill (6x15mm) is swallowed at 9 AM on day one. The recording is made until 4 PM and again from 8 AM until 2 PM on day two. The patient is placed in a bed and will be supplied with standardized food and fluid.

The Magnetic Tracking System consists of a 4 x 4 matrix of sensors positioned with respect to the anatomical reference points. Before measurements, the matrix is calibrated by offsetting the earth's and environmental magnetic fields. During the experiment, the magnet coordinates are continuously monitored and transmitted to a computer for processing and storage. Respiratory artifacts will be filtered out. Digestive movements will then be classified as 1) non-propulsive or 2) propulsive and transformed into either trajectory or dynamic graphs of the digestive motility.

The Magnetic Tracking System has the advantage from both radiographic and scintigraphic methods of conducting the tests without any radiation exposure to the patient. Preliminary studies have shown good concordance between the transit measured with the magnet and radiographic transit times.

The investigators wish to use this method, MTS, to compare the motility of the small intestine and the colon in patients with IBS-D and IBS-C as well as to compare these to groups to MTS done on healthy volunteers under the same conditions as the IBS patients.

DETAILED DESCRIPTION:
A MTS study on healthy volunteers is all ready done under the same conditions as described abow in Denmark. This study has projectID 20080037 and is approved by the Danish Dataprotection Agency as well as The Regional Committee on Biomedical Research Ethics.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18.
* Patients who are diagnosed with IBS according to the Rome III criteria.
* A total symptom score in GSRS-IBS at a minimum of 40 points.
* Patients who are psychologically stable and suitable for observation and able to provide informed consent.

Exclusion Criteria:

* Overt bowel diseases including inflammatory bowel disease.
* Pregnant or breast feeding.
* Patients who are considered unable to follow the planned programme of the study, including mental illness or physiological instability.
* Patients who are on medication with known influence on gastrointestinal motility including those for thyroid disease, diabetes mellitus, celiac disease and neurological disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 12 patients with IBS-D and 12 patients with IBS-C who all meet the inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2009-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janne Fassov, PhDstudent, Principal Investigator — Analfysiologisk Klinik, University Hospital of Aarhus
Locations (1):
- Analfysiologisk Klinik, University of Aarhus, Aarhus, Denmark